CLINICAL TRIAL: NCT06445192
Title: The BE FIT Study: Feasibility of an Exercise Intervention on Microbiome and Immune Function in a High-Risk Cohort for Lung Cancer
Brief Title: Evaluating the Impact of a Virtually Supervised Exercise Intervention and Group Counseling on Inflammation and the Microbiome of Smokers at High Risk for Lung Cancer, BE FIT Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Marisa Bittoni, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OSU-22194; NCI-2023-05556 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-10-17; First posted 2024-06-06 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Specimen Handling; Exercise Test; Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments will be obtained by research staff blinded to treatment group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (exercise intervention) (Experimental): Participants receive the supervised aerobic and resistance exercise intervention over 1 hour via telehealth BIW in weeks 1-8 and QW in weeks 9-12 and then continue with unsupervised exercise sessions BIW in weeks 13-52. Participants also attend group counseling sessions over 1 hour QW in weeks 1-8 and bi-weekly in weeks 9-12. Participants also wear a Fitbit throughout the trial and undergo collection of blood samples at baseline and follow up.
  Interventions: Procedure: Biospecimen Collection; Other: Exercise Counseling; Other: Exercise Intervention; Other: Medical Device Usage and Evaluation; Other: Physical Performance Testing; Other: Questionnaire Administration; Other: Telemedicine
- Group II (usual care) (Active Comparator): Participants receive usual care consisting of education on standard recommendations for physical activity, the benefits of exercise, and an example of a light walking program. Participants also wear a Fitbit throughout the trial and undergo collection of blood samples at baseline and follow up.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Other: Medical Device Usage and Evaluation; Other: Physical Performance Testing; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Group II (usual care)
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Exercise Counseling — Attend group counseling
  Arms: Group I (exercise intervention)
Other: Exercise Intervention — Receive aerobic and resistance exercise intervention via telehealth
  Arms: Group I (exercise intervention)
Other: Medical Device Usage and Evaluation — Wear Fitbit
Other: Physical Performance Testing — Ancillary studies
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Questionnaire Administration — Ancillary studies
Other: Telemedicine — Receive aerobic and resistance exercise intervention via telehealth
  Other Names: Telehealth
  Arms: Group I (exercise intervention)

SUMMARY:
This phase II trial evaluates how a virtually supervised exercise intervention in combination with group counseling affects inflammation and the bacterial composition (microbiome) of the gut in smokers who are at high risk for lung cancer. Physical exercise has been shown to reduce lung cancer development and to have beneficial effects on the gut microbiome and inflammation. Group counseling may promote adherence to the exercise intervention by empowering participants to exert greater control over their behavior and environment. This clinical trial may help researchers understand how exercise impacts inflammation and the microbiome in people at risk for lung cancer and whether or not exercise with counseling can improve health outcomes in high-risk individuals.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility and preliminary efficacy of establishing a multi-component virtually-delivered exercise intervention trial with longitudinal biomarker and microbiome collection in the Ohio State University Lung Cancer Screening Clinic (OSULCSC).

II. To determine the impact of the multi-component virtually-delivered exercise intervention on the microbiome and inflammatory biomarkers.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I: Participants receive the supervised aerobic and resistance exercise intervention over 1 hour via telehealth twice a week (BIW) in weeks 1-8 and once a week (QW) in weeks 9-12 and then continue with unsupervised exercise sessions BIW in weeks 13-52. Participants also attend group counseling sessions over 1 hour QW in weeks 1-8 and bi-weekly in weeks 9-12. Participants also wear a Fitbit throughout the trial and undergo collection of blood samples at baseline and follow up.

GROUP II: Participants receive usual care consisting of education on standard recommendations for physical activity, the benefits of exercise, and an example of a light walking program. Participants also wear a Fitbit throughout the trial and undergo collection of blood samples at baseline and follow up.

After completion of study intervention, participants are followed up at 12 weeks and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* 50-77 years of age
* Current or former smoker with 20-pack year smoking history and within the last 15 years
* Fewer than 150 minutes of participation in moderate intensity physical activity each week
* All participants must be free of severe heart, respiratory (e.g. chronic obstructive pulmonary disease [COPD]), or systemic disease that would make moderate intensity exercise participation unsafe
* Willing to sign an informed consent

Exclusion Criteria:

* Person undergoing treatment for cancer in any form
* Person plans to enter smoking cessation or change status

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients recruited to virtually-delivered exercise intervention (feasibility) | Up to 1 year
  To evaluate the feasibility and preliminary efficacy of establishing a multi-component virtually-delivered exercise intervention trial with longitudinal biomarker and microbiome collection in the Ohio State University Lung Cancer Screening Clinic (OSULCSC)
Proportion of patients who achieve study adherence (feasibility) based on attendance to the exercise program sessions and biospecimens submitted. | During 12-week program
  Study adherence is defined as a) the proportion of patients attending at least 20 out of 24 sessions for the 12-week program and b) the percentage of biospecimen samples collected at the post program period (12 weeks). This study will be considered feasible if the compliance rate for both of these combined is 75% or more. Descriptive statistics will be used to examine the distribution of all patient and treatment characteristics, including compliance.
Assess the number of participants with a change in inflammatory biomarkers | Baseline to post-intervention (12 weeks)
  Will assess the effect of the intervention on inflammatory markers of C-reactive protein and IL-6 separately using linear mixed models with the biomarker serving as the outcome variable. Will also assess the changes in the biomarkers across time in each intervention group.
Microbe relative abundances | Baseline to post-intervention (12 weeks)
  Will assess the effect of the intervention on the diversity and relative abundances of individual microbes. Will compare everyone's post-intervention time point to baseline in control and the exercise interventions cohorts, applying linear or generalized mixed-effects models for the diversity or individual microbes.

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Bittoni, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu